CLINICAL TRIAL: NCT01842646
Title: A Phase II Study Evaluating the Oral Smoothened Inhibitor PF-04449913 in Patients With Myelodysplastic Syndrome (MDS)
Brief Title: Phase II Hedgehog Inhibitor for Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17302
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Results first posted 2017-03-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Myelodysplastic Syndrome (MDS); Chronic Myelomonocytic Leukemia (CMML)
Keywords: Leukemia; Myeloid Malignancies
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia | interventions — glasdegib; SMO protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-04449913 Treatment (Experimental): Treatment will be administered on an outpatient basis. All patients will be treated with an oral dose PF-04449913 at 100 mg daily in 4-week cycles for a total of 4 cycles. Patients who demonstrate no evidence of progressive disease (i.e. stable disease or better) may continue on treatment until disease progression or loss of response, limiting toxicity, or death.
  Interventions: Drug: PF-04449913

INTERVENTIONS:
Drug: PF-04449913 — Patients will be enrolled according to a two-step study design. Twenty patients will be enrolled in the first stage. All patients will be given a daily oral dose of PF-0444913 100 mg for up to 4 cycles, with an optional continuation phase. Dose escalation to 200 mg will be provided for patients who do not have at least hematologic improvement following 2 cycles, and dose reduction to 50 mg will be permitted for patients with significant toxicity. If at least 2 patients respond in the initial stage, and additional 15 patients will be enrolled in the second stage.
  Other Names: Oral Hedgehog Inhibitor; Smoothened (SMO) Inhibitor

SUMMARY:
This study is being done to see how safe an investigational drug is and test how well it will work to help people with refractory/relapsed myelodysplastic syndrome (MDS) or chronic myelomonocytic leukemia (CMML).

DETAILED DESCRIPTION:
The main purpose of this study is to see whether the participant's disease responds favorably to the investigational drug, PF-04449913.

Post treatment Phase: After coming off of active treatment study drug (PF-04449913), participants will be followed monthly for survival only. No other data will be captured during this time.

ELIGIBILITY:
Inclusion Criteria:

* Must have a pathologically confirmed diagnosis by World Health Organization (WHO) Criteria of MDS, CMML, or acute myeloid leukemia (AML) (except acute promyelocytic leukemia) with < 30% bone marrow blasts (RAEB-t by French American British criteria)
* Hypomethylating agent (azacitidine and/or decitabine) failure, defined as lack of response, disease progression, loss of response, or intolerance as deemed by the study investigator
* Adequate renal function, as evidenced by a serum creatinine ≤ 2 times the institutional upper limit of normal
* Adequate hepatic function, as evidenced by a serum bilirubin < 2 times the institutional upper limit of normal and an aspartic transaminase (AST) and alanine transaminase (ALT) < 2 times the institutional upper limit of normal. Indirect hyperbilirubinemia due to Gilbert's disease or hemolysis is permitted.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with a history of prior therapy with another investigational agent within 4 weeks of the first planned dose of PF-0444913
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PF-04449913
* Prior therapy with another hedgehog inhibitor
* Concurrent use of any other agent for MDS, CMML, or AML. Growth factor use with epoetin, darbepoetin, or granulocyte colony-stimulating factor must be terminated at least 2 weeks before initiation of study treatment.
* Any uncontrolled concurrent illness that would, in the opinion of the investigator, limit compliance with study requirements
* Second malignancy requiring active therapy
* A prolonged corrected QT interval (QTc) of ≥480 ms interval on electrocardiogram
* History of metastatic cancer diagnosed less than 2 years prior to the first planned dose of PF-0444913
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because PF-04449913 is smoothened inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with PF-04449913. Breastfeeding should be discontinued if the mother is treated with PF-04449913.
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination antiretroviral therapy are excluded from the study because of possible pharmacokinetic interactions with PF-04449913.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-08-29 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Lancet, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in August 2013 and participants were enrolled at Moffitt Cancer Center between September 2013 and September 2015.
Groups:
- Experimental: PF-04449913 Treatment: Treatment to be administered on an outpatient basis. All participants to be treated with an oral dose PF-04449913 at 100 mg daily in 4-week cycles for a total of 4 cycles.
Period: Overall Study
Arm/Group | Experimental: PF-04449913 Treatment
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Experimental: PF-04449913 Treatment
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 29
Age, Continuous [Median (Full Range); unit: years] | 75 [55 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall International Working Group (IWG) 2006 Response Rate
Description: Response recorded from the start of the treatment until disease progression/recurrence. All responses must last for at least 8 weeks. Complete Remission (CR): Bone marrow: ≤ 5% myeloblasts with normal maturation of all cell lines, Persistent dysplasia will be noted, Peripheral blood: Hemoglobin ≥ 11 g/dL, Platelets ≥ 100 x 10^9/L, Neutrophils ≥ 1.0 x 10^9/L, Blasts 0% ; Partial Remission (PR): All CR criteria if abnormal before treatment, except: Bone marrow blasts decreased by ≥ 50% over pretreatment but still > 5%, Cellularity and morphology not relevant; Marrow CR or Hematological Improvement (HI): Bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment Peripheral blood: if HI responses, they will be noted in addition to marrow CR. Further investigation of PF-04449913 would not be warranted if it produced an overall response rate (CR + PR + marrow CR+HI) of 10% or less (p0), and would be warranted if it produced an overall response rate of 30% or more (p1).
Time Frame: Up to 2 years, 4 months
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: PF-04449913 Treatment
Number analyzed (Participants) | 35
Participants
  Complete Remission (CR) | 0
  Hematological Improvement (HI) | 2
  Stable Disease (SD) | 19
  Progressive Disease (PD) | 14

2. Secondary Outcome: Median Overall Survival (OS)
Description: To estimate the overall survival of patients with refractory/relapsed myelodysplastic Syndrome (MDS) and chronic myelo-monocytic leukemia (CMML) treated with PF-0444913. Overall survival will be defined as the time period between the date of the first dose of drug until the time of death.
Time Frame: Up to 2 years, 4 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: PF-04449913 Treatment
Number analyzed (Participants) | 35
months | 10.2 [6.8 to 13.6]

3. Secondary Outcome: Median Event Free Survival
Description: To estimate the event-free survival of patients of this population. Event-free survival will be defined as the date of the first dose of study drug until failure (disease progression) or death from any cause.
Time Frame: Up to 2 years, 4 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: PF-04449913 Treatment
Number analyzed (Participants) | 35
months | 6.4 [1.9 to 18.33]

4. Secondary Outcome: Median Time to Transformation to Acute Myeloid Leukemia (AML)
Description: To estimate the time to transformation to AML in patients with <20% blasts. In patients with less than 20% blasts, the time to transformation to AML will be defined as the date of the first dose of drug until either the percentage of bone marrow blasts or the percentage of peripheral blasts exceeds 20%, whichever is first.
Time Frame: Up to 2 years, 4 months
Population: NA- The median time to AML was not reached due to insufficient number of participants with events.
Arm/Group | Experimental: PF-04449913 Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment emergent adverse events occurring in equal to or more than 10% of participants.
Time Frame: 2 years, 4 months
Population: All participants
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: PF-04449913 Treatment
Number analyzed (Participants) | 35
Participants
  Grade 1-2 : Pain | 22
  Grade 1-2 : Dysgeusia | 21
  Grade 1-2 : Nausea | 11
  Grade 1-2 : Anorexia | 11
  Grade 1-2 : Skin/rash | 8
  Grade 1-2 : Oral mucositis | 9
  Grade 1-2 : AST elevated | 8
  Grade 1-2 : Alopecia | 8
  Grade 1-2 : ALT elevated | 6
  Grade 1-2 : Dizziness | 6
  Grade 1-2 : Dyspnea | 5
  Grade 1-2 : Infections | 2
  Grade 1-2 : Fatigue | 6
  Grade 1-2 : Diarrhea | 6
  Grade 1-2 : Constipation | 5
  Grade 1-2 : Fever | 5
  Grade 1-2 : Hyperkalemia | 5
  Grade 1-2 : Hyperglycemia | 4
  Grade 1-2 : Thrombocytopenia | 2
  Grade 1-2 : Headache | 4
  Grade 1-2 : Vomiting | 4
  Grade 3-4 : Pain | 1
  Grade 3-4 : Dysgeusia | 0
  Grade 3-4 : Nausea | 0
  Grade 3-4 : Anorexia | 0
  Grade 3-4 : Skin/rash | 1
  Grade 3-4 : Oral mucositis | 0
  Grade 3-4 : AST elevated | 0
  Grade 3-4 : Alopecia | 0
  Grade 3-4 : ALT elevated | 0
  Grade 3-4 : Dizziness | 0
  Grade 3-4 : Dyspnea | 1
  Grade 3-4 : Infections | 4
  Grade 3-4 : Fatigue | 0
  Grade 3-4 : Diarrhea | 0
  Grade 3-4 : Constipation | 0
  Grade 3-4 : Fever | 0
  Grade 3-4 : Hyperkalemia | 0
  Grade 3-4 : Hyperglycemia | 0
  Grade 3-4 : Thrombocytopenia | 2
  Grade 3-4 : Headache | 0
  Grade 3-4 : Vomiting | 0

ADVERSE EVENTS:
Time Frame: 2 years, 4 months
Arm/Group | Experimental: PF-04449913 Treatment
Serious Adverse Events (participants affected / at risk) | 11/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: PF-04449913 Treatment (N=35)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (2)
Death NOS (General disorders) | 2 (2)
Abdominal infection (Infections and infestations) | 1 (1)
Bone infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, GI (Infections and infestations) | 1 (1)
Infections and infestations - Other, Rhinovirus/Enterovirus (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, possible DLBCL NHL (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: PF-04449913 Treatment (N=35)
Pain (General disorders) | 23 (30)
Fatigue (General disorders) | 6 (6)
Fever (General disorders) | 5 (5)
Edema limbs (General disorders) | 3 (3)
Flu like symptoms (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
General disorders and administration site conditions - Other (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 21 (25)
Dizziness (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 4 (5)
Memory impairment (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Dysarthria (Nervous system disorders) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (9)
Alanine aminotransferase increased (Investigations) | 6 (10)
Weight loss (Investigations) | 5 (5)
Platelet count decreased (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 2 (2)
Neutrophil count decreased (Investigations) | 2 (2)
Investigations - Other (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 11 (14)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (4)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 11 (13)
Mucositis oral (Gastrointestinal disorders) | 9 (9)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 4 (7)
Skin infection (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (3)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Testicular hemorrhage (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes